CLINICAL TRIAL: NCT03123419
Title: Gardasil Administration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Departmental research hold
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Sarah Hostetter, MD, Principal Investigator, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 27734
Record Dates: First submitted 2017-04-10; First posted 2017-04-21 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Vaccine Administration Rates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaccine (Other): All patients who consent to be in the study will receive Appointment reminders.
  Interventions: Behavioral: Appointment reminders

INTERVENTIONS:
Behavioral: Appointment reminders — The purpose of the Gardasil study is to increase the rates of Gardasil vaccination in the Maternal Fetal Care Center. This will be done by reminding patients via text to come for their follow up vaccine appointments.

SUMMARY:
The purpose of the Gardasil study is to increase the rates of Gardasil vaccination at a maternal fetal Care Center. This will be done by reminding patients via text to come for follow up vaccine appointments.

DETAILED DESCRIPTION:
Patients will be screened in center for history of Gardasil vaccination. If the patient has not received the vaccination series they will be counseled/educated (standard of care [SOC }) and offered the vaccine series. If the patient agrees to the vaccination, they will then be offered participation in this study, (consent will be reviewed and signed) and they will receive the first vaccination at this visit, administered according to standard protocol. The patient will then be scheduled for two follow up vaccination appointments. The second vaccination will be given 2 months after the first vaccine and the third will be given 4 months after the second vaccination in accordance with the Gardasil vaccine guidelines. -SOC

The patients will receive a total of two texts during the study entirety. The two texts will be appointment reminders for the second and third vaccination, sent 1 week prior to the next appointment. This is study related.

Data collection Data will be collected using a data collection sheet. The investigators will record date of first vaccine administration and adherence to follow up.vaccinations.

ELIGIBILITY:
Inclusion criteria

* Patient receiving gynecological or postpartum care at the Maternal Fetal Care Center
* Females age 9-26 years per manufacturer's recommendation
* Having a cell phone that will allow texting
* Willing to accept any texting charges that may occur for receiving the reminder text.

Exclusion criteria

* Allergy to HPV-4 or HPV-9 vaccine
* Prior completion of the HPV-4/9 series,
* Pregnancy
* Patients older than 26 years old

Ages: 9 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Increase HPV-9 vaccine administration rates | through study completion, an average of 1 year
  The text reminder messages will increase HPV-9 vaccine administration rates

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hostetter, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No